CLINICAL TRIAL: NCT07006454
Title: Comparison of Ventro-Cephalic to Dorso-Caudal Translatoric Glides in Management of Cervicogenic Headache
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/79
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-16 (Actual); Status verified 2024-07

CONDITIONS: Cervicogenic Headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Participants of group A will receive ventro-cephalic translatoric glide, total of 3 sets with 15 repetitions per set.
  Duration (5 treatment sessions per week for 2 weeks)
  Interventions: Procedure: Ventro-Cephalic Translatoric Glide
- Group B (Experimental): Participants of group B will receive Dorso-caudal translatoric glide, total of 3 sets with 15 repetitions per set.
  Duration (5 treatment sessions per week for 2 weeks)
  Interventions: Procedure: Dorso-Caudal Translatoric Glide

INTERVENTIONS:
Procedure: Ventro-Cephalic Translatoric Glide — Participants of group A will receive ventro-cephalic translatoric glides, total of 3 sets with 15 repetitions per set.
  PROCEDURE:
  1. Patient sits on low chair with back straight and therapist stand facing the patient's right side.
  2. Therapist's stable hand: with the thumb and index finger of left hand fixate caudal vertebra.
  3. Therapist's moving hand: therapist will place his/her right hand on left side of patient's head and cervical spine than place little finger around cranial vertebra of segment to be moved.
  4. Apply glide in ventro-cranial direction in the right angle of the treatment plane of the facet joint.
  Arms: Group A
Procedure: Dorso-Caudal Translatoric Glide — Participants of group B will receive Dorso-caudal translatoric glides, total of 3 sets with 15 repetitions per set.
  PROCEDURE:
  1. Patient sits on low chair with back straight and therapist stand facing the patient's left side.
  2. Therapist's stable hand: with the thumb and index finger of right hand fixate caudal vertebra.
  3. Therapist's moving hand: therapist will place his/her left hand on right side of patient's head and cervical spine than place little finger around cranial vertebra of segment to be moved.
  4. Apply glide in dorso-caudal direction in the right angle of the treatment plane of the facet joint.
  Arms: Group B

SUMMARY:
This study is a randomised control trial and the purpose of this study is to compare ventro-cephalic to dorso-caudal translatoric glides in management of cervicogenic headache.

DETAILED DESCRIPTION:
Participants will be recruited into their respective groups using a coin toss method.Cervicogenic headache will be assesed using International Classification of Headache Disorders, 3rd edition:

A- Any headache fulling criterion C. B- Clinical and/or imaging evidence of lesion or disorder in cervical spine or soft tissues of neck that can cause headache.

C- Evidence of cause of headache demonstrated by at least 2 of these:

1. headache has developed in temporal relation to the onset of the cervical disorder or lesion.
2. headache has significantly improved or resolved in parallel with improvement in cervical lesion or disorder.
3. cervical range of motion is reduced, and headache is made significantly worse by provocative maneuvers.
4. headache is abolished following anaesthetic blocked of cervical structure. D- Not better accounted for by another ICHD-3 diagnosis.

CEH subject selection is based on clinical criteria, however anaesthetic blockades is not used as a criterion.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18 to 44 years old

  * Both male and female A- Any headache fulling criterion C. B- Clinical and/or imaging evidence of lesion or disorder in cervical spine or soft tissues of neck that can cause headache.

C- Evidence of cause of headache demonstrated by at least 2 of these:

1. headache has developed in temporal relation to the onset of the cervical disorder or lesion.
2. headache has significantly improved or resolved in parallel with improvement in cervical lesion or disorder.
3. cervical range of motion is reduced, and headache is made significantly worse by provocative maneuvers.
4. headache is abolished following diagnostic blocked of cervical structure. D- Not better accounted for by another ICHD-3 diagnosis

Exclusion Criteria:

* 1- Tension-type headaches and migraine 2- History of Vertigo or Dizziness 3- Already taking manual therapy treatment 4- Prior surgery to the head and neck 5- Trauma

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Headache intensity | Variable will be evaluated at baseline and then weekly for next 2 weeks.
  It will be measured on a numeric pain rating scale where participant select number ranging from 0 to 10 based on pain intensity, with 0 representing no pain and 10 denotes extreme pain.
Headache disability | Variable will be evaluated at baseline and then weekly for next 2 weeks
  It will be measured using headache disability index (HDI) which is a 25 item self-rated questionnaire in which participants rate their headache disability by selecting an option from 1 to 3 (yes= 4 points, sometimes= 2 points, and No = 0 point) then sum of responses is used to get final score.
  Interpretation:
  10 to 28= mild disability 30 to 48= moderate disability 50 to 68= severe disability 72 or more= complete disability
Quality of Life of patient | Variable will be evaluated at baseline and then weekly for next 2 weeks
  It will be measured using headache impact test (HIT-6), this tool is used to measure impact of headache on ability to function, a 6 items self-rated questionnaire in which participant select an option from 1 to 5 (Never= 6 points, rarely= 8, sometimes= 10, very often= 11, always= 13) then sum of responses is used to get final score.
  Interpretation:
  60 or more= Very severe impact 56 to 59= Substantial impact 50 to 55= Some impact 49 or less= Little or no impact
Headache Frequency | Variable will be evaluated at baseline and then weekly for next 2 weeks
  It will be measured using medical diary, which is a self-reported measure in which the patient will be asked to report the number of headache days per week through a medical logbook, which will be recorded every day and night.
Cervical range of motion | Variable will be evaluated at baseline and then weekly for next 2 weeks
  It will be measured using CROM instrument a plastic frame device that is fastened to the head with help of Velcro-strap, it consist of 3 separate inclinometers that are fixed to frame (1 in sagittal plan which evaluates range of motion in flexion and extension, where 2nd in frontal plane which evaluates range of motion in side bending, and 3rd in horizontal plan which indicates range of motion in rotation)
Cervical flexion rotation test | Variable will be evaluated at baseline and then weekly for next 2 weeks
  It is used to evaluate impairment of cervical function as the diagnostic criterion of internation headache society (IHS) consist of subjective feathers which includes impairments at atlanto-axial motion segments which is assessed by cervical flexion rotation test.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan